CLINICAL TRIAL: NCT02386722
Title: Impact of a Pharmaceutical Care Intervention to Improve Adherence of Inhaled Medication in Asthma and COPD Patients
Brief Title: Intervention to Improve Inhalative Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hosptal, Baselland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jörg Leuppi, Head University Clinic of Internal Medicine, Canton Hospital Baselland, Cantonal Hosptal, Baselland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 269/13
Record Dates: First submitted 2014-02-14; First posted 2015-03-12 (Estimated); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Chronic Asthma; COPD
Keywords: Adherence of inhaled medication; pharmaceutical intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention group (Experimental): The intervention consisted of an audio-reminder, generated by an app (in case of SmartInhaler devices) or in form of an alarm clock (for the POEMS), and directly transferred to the participants' smartphones. Patients were allowed to choose the inhalation times themselves. The reminder generated by the by the smartphone had to be quitted by the patients. Patients in the intervention group received support calls carried out by the pharmacist or trained study nurses, when the use of rescue medication doubled or when the medication was not inhaled as prescribed for more than two consecutive days. Participants also received a feedback on their adherence at each clinical visit, especially for the results of the POEMS.
  Interventions: Device: Electronic Monitoring with audio reminders and additional support
- Control group (No Intervention): Patients in the control group received a Smartinhaler/POEMS, which only records their adherence. Patients assigned to the control group did not receive any reminder or support regarding their adherence to inhaled medication.

INTERVENTIONS:
Device: Electronic Monitoring with audio reminders and additional support — Automated reminder:
  -Daily audio-reminder, generated by a smartphone.
  Support calls (only patients with Smartinhaler):
  * When the use of rescue medication doubles.
  * When inhaled medication was not inhaled as prescribed for more than two consecutive days.
  Feedback on adherence (only patients with POEMS):
  -At every clinical visit (after 2, 4 and 6 months).
  Arms: Intervention group

SUMMARY:
Despite progress in pharmacological and non-pharmacological treatment in recent years, the burden of disease among asthma and COPD patients is high and patients may be frequently hospitalized due to exacerbations. Reasons for uncontrolled disease are manifold, but are frequently associated with poor inhalation technique and non-adherence to the prescribed treatment plan which may cause substantial mortality, morbidity, and cost to the healthcare system. In this respect, the study of causes for non-adherence and the development of measures to increase respectively maintain treatment adherence, particularly in chronic diseases, is of major clinical importance.

The aim of this study was to investigate the impact of an acoustic reminder and a close supervision on adherence to inhaled medication and on course of disease and quality of life (Qol) in asthma and COPD patients.

In this single-blinded trial, asthma and/or COPD patients were randomly assigned either to the intervention or the control group. Adherence to inhaled medication was monitored using electronic data capture devices, recording date and time of each inhalation device actuation. Follow-up was six months. Primary outcome was defined as "time to next exacerbation". Secondary outcomes included number of exacerbations, number of exacerbations with hospitalization, taking/timing adherence, and Qol during follow-up. Adherence was measured using electronic data capture devices which saved date and time of each inhalative device actuation. Patients are randomly assigned to an intervention, respectively control group. Patients assigned to the intervention group will receive audio reminder and support calls in case medication is not been taken as prescribed or if rescue medication is used more frequently than prespecified in the study protocol. During the study, participants are assessed every two months.

ELIGIBILITY:
Inclusion:

* Aged 18 years or older
* Have an established asthma-diagnosis according to the Global Initiative for Asthma (GINA) guidelines and/or
* Have an established COPD diagnosis according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (severity GOLD I-IV based on the international GOLD-Criteria) [46] and
* Are prescribed daily inhaled medication (controller medication for a daily maintenance treatment)
* Had at least one exacerbation in the previous 12 months before study start
* With a metered dose Inhaler (e.g. Ventolin®), Diskus (e.g.Seretide®), Turbohaler (e.g.Symbicort®), Aerolizer/Breezhaler (e.g.Onbrez®), HandiHaler (e.g. Spiriva®) or Ellipta (e.g Relvar®)

Exclusion:

* Suffering from malignancies and/or other severe diseases
* Insufficient in the German language
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Leuppi, Prof.MD PhD, Principal Investigator — 061 925 21 81
Locations (2):
- Switzerland (2):
  - Cantonal Hospital Baselland Liestal, Liestal, Basel-Landschaft
  - Cantonal Hospital Baselland, Liestal, Basel-Landschaft

REFERENCES:
- [Derived] Gregoriano C, Dieterle T, Breitenstein AL, Durr S, Baum A, Giezendanner S, Maier S, Leuppi-Taegtmeyer A, Arnet I, Hersberger KE, Leuppi JD. Does a tailored intervention to promote adherence in patients with chronic lung disease affect exacerbations? A randomized controlled trial. Respir Res. 2019 Dec 3;20(1):273. doi: 10.1186/s12931-019-1219-3. PMID 31796013
- [Derived] Gregoriano C, Dieterle T, Durr S, Arnet I, Hersberger KE, Leuppi JD. Impact of an Electronic Monitoring Intervention to Improve Adherence to Inhaled Medication in Patients with Asthma and Chronic Obstructive Pulmonary Disease: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Oct 23;6(10):e204. doi: 10.2196/resprot.7522. PMID 29061556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from several hospitals in the Basel region and patients treated by pulmonologists in private practice are screened for eligibility. In addition, advertisement is made using posters, flyers, as well as on ad-screens. Advertisement is also placed in local newspapers.
  Enrolment started on January 2014 and will ended on September 2017.
Pre-assignment Details: Prior to randomization, all participants take part in a training course before the baseline visit. The goal of the training course is to provide refresher training on inhalation techniques in order to ensure that all participants are at the same level of disease knowledge and use their medication correctly.
Groups:
- Intervention Group: The intervention consisted of an audio-reminder, generated by an app (in case of SmartInhaler devices) or in form of an alarm clock (for the POEMS), and directly transferred to the participant's smartphones. In addition, patients in the intervention group received support calls carried out by the pharmacist, when the use of rescue medication doubled respectively when the inhaled medication was not inhaled as prescribed for more than two consecutive days. Participants also received a feedback from the pharmacist on their adherence at each clinical visit, especially for the results of the POEMS.
- Control Group: Patients in the control group received a Smartinhaler/POEMS, which only records their adherence. The alarm function of the devices will be switched off, and these participants will not be reminded to take their inhalers. This group will not receive any calls, if they do not comply with the prescribed medication schedule or if they use their rescue medication too frequently.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started (4 Patients withdrew consent prior to randomization, so that only 165 patients were randomized.) | 84 | 81
Completed | 75 | 74
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Patients were randomly assigned either to the intervention or control group. The intervention consisted of an audio-reminder, generated by an app (in case of SmartInhaler devices) or in form of an alarm clock (for the POEMS), and directly transferred to the participant's smartphones. In addition, patients in the intervention group received support calls carried out by the pharmacist, when the use of rescue medication doubled respectively when the inhaled medication was not inhaled as prescribed for more than two consecutive days. Participants also received a feedback from the pharmacist on their adherence at each clinical visit, especially for the results of the POEMS.
  Smartinhaler/POEMS with audio reminders and additional support calls: Patients assigned to the intervention group will receive a Smartinhaler/POEMS, which will contain an audio reminder function. If the alarm function is on, a ring tone will be generated, after the time predesigned for inhalation. If the use of
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.8) | 64.7 (12.4) | 68.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 52
  Male | 51 | 46 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Next Asthma or COPD Exacerbation up to 182 Days
Description: The primary outcome of this study was "time to next asthma or COPD exacerbation", defined as acute-onset worsening of the patient's condition beyond day-to-day variations requiring interaction with a healthcare provider. It was expressed as the number of exacerbations since the last visit with the exact period of exacerbation also including the number of exacerbations requiring hospitalisation. The first exacerbations during the study period served as reference to calculate the primary endpoint "time to next exacerbation".
Time Frame: 182 days
Measure: Mean (Full Range); unit: days to first exacerbation
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 75 | 74
days to first exacerbation | 172 [161 to 182] | 161 [149 to 174]

2. Secondary Outcome: Number of Exacerbations.
Description: Number of exacerbations during the study period.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: number of exacerbations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 75 | 74
number of exacerbations | 0.3 (0.6) | 0.5 (1.0)

3. Secondary Outcome: Number of Severe Exacerbations.
Description: Exacerbations with the need for hospitalization.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: severe exacerbations
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 75 | 74
severe exacerbations | 0.08 (0.3) | 0.08 (0.4)

4. Secondary Outcome: Adherence to Puff Inhalers
Description: Mean duration with Adherence to Puff Inhalers in the Target Range
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: days in target range
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 57 | 60
days in target range | 81.6 (14.2) | 60.1 (30.3)

5. Secondary Outcome: Percentage of Days With Adherence to Dry Powder Capsules (Breezhaler and Handihaler) Assessed by POEMS
Description: percentage of days with Adherence to Dry Powder Capsules. Taking adherence = [number of puffs inhaled during 24 hours / number of puffs prescribed during 24 hours) x 100. Correct taking adherence was considered when taking adherence was between 80-100%, based on previous studies.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: % of days in target range
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 49
% of days in target range | 89.6 (9.8) | 80.2 (21.3)

6. Secondary Outcome: Percentage of Days of Adherence
Description: percentage of days of Adherence for puff inhalers (metered dose inhalers, Turbohaler, Discus, Ellipta) assessed by Smartinhalers.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: % of days in target range
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 57 | 60
% of days in target range | 68.9 (25.0) | 50.6 (32.5)

7. Secondary Outcome: Percentage of Days With Timing Adherence
Description: percentage of days with timing Adherence for dry powder capsules (Breezhaler, Handihaler), assessed by POEMS
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: % of days in target range
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 49
% of days in target range | 79.6 (12.9) | 71.7 (22.0)

8. Secondary Outcome: Percentage of Gaps in Puff Inhaler Use
Description: Percentage of Gaps in Puff Inhaler Use Gaps = [number of days without inhalation during the whole study period / number of days in same time period] x 100.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: % of gaps
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 57 | 60
% of gaps | 3.2 (4.7) | 11.7 (18.6)

9. Secondary Outcome: Percentage of Gaps for Dry Powder Capsules (Breezhaler, Handihaler), Assessed by POEMS.
Description: Percentage of Gaps = [number of days without inhalation during the whole study period / number of days in same time period]
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: % gaps
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 49
% gaps | 4.6 (4.4) | 9.8 (8.9)

10. Secondary Outcome: Numbers of Days of the Longest Period of Time Without Inhalation During the Investigated Time Period
Description: Maximal gap length = number of consecutive days of the longest period of time without Inhalation during the investigated timeperiod.Assessed by Smartinhalers.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 57 | 60
days | 1.6 (2.0) | 11.6 (25.6)

11. Secondary Outcome: Number of Days of the Longest Period of Time Without Inhalation.
Description: Maximal gap length for dry powder capsules (Breezhaler, Handihaler), Assessed by POEMS = number of consecutive days of the longest period of time without inhalation.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 49
days | 2.6 (2.7) | 5.9 (5.2)

12. Secondary Outcome: Score of the St. George Respiratory Questionnaire
Description: Score of the St. George Respiratory Questionnaire. Quality of life was assessed using the St. George Respiratory Questionnaire. This is a questionnaire, which was developed for measuring impaired health and perceived well-being in patients with asthma and COPD. Each Subscore ranges from 0-100, higher scores indicate more limitations in one of the 4 domains.
  Subscore Symptoms (ranges from 0-100): higher scores indicate worse outcome Subscore Activity (ranges from 0-100): higher scores indicate worse outcome Subscore Impact (ranges from 0-100): higher scores indicate worse outcome
  Total Score (ranges from 0-100): higher scores indicate worse outcome. The total score is calculated as a weighted sum of the three subscores. Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 75 | 74
score on a scale
  Subscore Symptoms | 45.7 (21.5) | 48.7 (25.6)
  Subscore Activity | 45.2 (19.3) | 52.4 (23.7)
  Subscore Impact | 21.8 (14.6) | 29.3 (20.7)
  Total Score | 32.5 (14.7) | 39.6 (20.3)

ADVERSE EVENTS:
Time Frame: Study duration of 6 months
Description: All participants have the same minimal risk for adverse events not related to the study.
  Patients were not exposed to any risk by participating in this study. Patients continued to use their prescribed medication as usual. Study participants were cared for by their usual physician(s). The diagnostic tests were carried out at low risk.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/81
Other Adverse Events (participants affected / at risk) | 0/84 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02386722/Prot_SAP_000.pdf